CLINICAL TRIAL: NCT01212159
Title: Telephone Based Management of Hyperlipidemia Utilizing a Self Monitoring Testing Device
Brief Title: Telephone Based Management of Hyperlipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alfred A Bove, MD, PhD, Emeritus Professor of Medicine, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12832
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Hyperlipidemia
Keywords: Internet based monitoring system
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No self monitoring device (No Intervention): Standard or usual care of high LDL including lab lipid profiles after treatment with statin therapy. No device or telemedicine education will be provided
- Self Monitoring Lipid Analyzer (Experimental): Self measured blood lipids using a home lipidometer, and telephone reporting of data to the clinical center.
  Interventions: Device: Self Monitoring Lipid Analyzer

INTERVENTIONS:
Device: Self Monitoring Lipid Analyzer — The device is similar to a glucometer- Utilizing a lancet a small amount of blood is collected in a capillary tube and placed on a hand held monitor that records lipid values.
  Other Names: Cardiochek
  Arms: Self Monitoring Lipid Analyzer

SUMMARY:
The purpose of the study is to demonstrate that systematic self measurement of blood lipids reduces LDL cholesterol more effectively than standard care. The hypothesis is that cholesterol lowering medication adherence will be improved with self monitoring and reporting of frequent blood lipids and the percentage of patients achieving LDL goal will be greater than without home monitoring.

DETAILED DESCRIPTION:
The study utilizes a telephone reporting system to self report lipid values and provide educational counseling regarding lifestyle modification methods to reduce cardiovascular risk. Study patients will be randomized to receive a home monitoring device and will be instructed on its use. Generic simvastatin will be given to reduce LDL levels in all groups. It is the hypothesis that those study patients receiving a home device will reach target LDL (goal LDL) more frequently than those randomized to usual care( no device).

ELIGIBILITY:
Inclusion Criteria:

* LDL > 130mg/dl

Exclusion Criteria:

* Pregnant patients
* liver disease
* allergic reaction to statins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Self Monitoring Device | Self Monitoring Lipid Analyzer
Started | 26 | 44
Completed | 14 | 32
Not Completed | 12 | 12
Not completed — Withdrawal by Subject | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Self Monitoring Device | Self Monitoring Lipid Analyzer | Total
Number analyzed (Participants) | 14 | 32 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.6) | 52.5 (9.3) | 54.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 27 | 33
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 28 | 29
  Not Hispanic or Latino | 12 | 3 | 15
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 19 | 26
  White | 5 | 9 | 14
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 32 | 46

OUTCOME MEASURES:

1. Primary Outcome: LDL Level Change From Baseline
Description: Comparison of serum LDL level between control and intervention subjects
Time Frame: baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | No Self Monitoring Device | Self Monitoring Lipid Analyzer
Number analyzed (Participants) | 14 | 32
mg/dl | -63.4 (35.5) | -54.6 (43.2)
Statistical Analysis 1: Comparison: No Self Monitoring Device vs Self Monitoring Lipid Analyzer; Paired t-test analysis of 6 month change in LDL cholesterol for no monitor and self monitor groups Independent sample t-test to compare ldl change between groups; Test type: Superiority or Other; p = 0.391, t-test, 2 sided — Comparison of mean reduction in LDL cholesterol between no monitor (control) and monitor (intervention) groups

2. Secondary Outcome: Medication Compliance
Description: Self reported comparison of lipid medication compliance between control and intervention subjects, scale 0-4. Highest compliance value indicated by a score of 4.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Self Monitoring Device | Self Monitoring Lipid Analyzer
Number analyzed (Participants) | 14 | 32
units on a scale | 2.4 (1.1) | 2.4 (1.2)

3. Secondary Outcome: LDL Values at Two Week Interval
Description: Participant in the self monitored arm reported LDL every two weeks. LDL goal for treatment was 100 mg/dl and subjects were followed every two weeks to observe mean LDL values.
Time Frame: 6 weeks
Population: No self monitoring group had LDL levels only at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | No Self Monitoring Device | Self Monitoring Lipid Analyzer
Number analyzed (Participants) | 0 | 32
mg/dl
  two week |  | 96.3 (47.3)
  four week |  | 92.4 (37.0)
  six week |  | 118.6 (37.8)

ADVERSE EVENTS:
Arm/Group | No Self Monitoring Device | Self Monitoring Lipid Analyzer
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/44
Other Adverse Events (participants affected / at risk) | 0/26 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Self Monitoring Device (N=26) | Self Monitoring Lipid Analyzer (N=44)
Motor vehicle accident, minor musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject seen in emergency department after MVA, analgesic therapy prescribed for 4 days.
Hodgkins lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Subject noted to have lymphadenopathy during study period. Evaluation by hematology diagnosed Hodgkin's lymphoma and instituted therapy. Subject withdrew from study before completion.

LIMITATIONS AND CAVEATS:
Recruiting did not reach goal due to change in FDA approval for simvastatin use requiring protocol modification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No